CLINICAL TRIAL: NCT03824223
Title: 'Fitness To Fly' Testing In Children With Neuromuscular Weakness Or Central Hypoventilation: A Feasibility Study
Brief Title: 'Fitness To Fly' Tests In Children With Type II Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Collaborators: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 17IA16
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-12

CONDITIONS: Neuromuscular Diseases; Central Hypoventilation
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Intervention Model Description: Participants randomised to uniform balanced crossover (new/old or old/new hypoxic challenge test components).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- new/old HCT component order (Other): new/old hypoxic challenge test (HCT) component order
  Where the new test uses pulse oximetry and transcutaneous CO2 monitoring to guide use of ventilatory support and if necessary supplementary oxygen and the old test uses pulse oximetry to titrate supplementary oxygen.
  Interventions: Diagnostic Test: Hypoxic challenge test
- old/new HCT component order (Other): old/new hypoxic challenge test (HCT) component order
  Where the old test uses pulse oximetry to titrate supplementary oxygen and the new test uses pulse oximetry and transcutaneous CO2 monitoring to guide use of ventilatory support and if necessary supplementary oxygen.
  Interventions: Diagnostic Test: Hypoxic challenge test

INTERVENTIONS:
Diagnostic Test: Hypoxic challenge test — Physiological response to 15% ambient oxygen monitored.

SUMMARY:
The conventional hypoxic challenge test might not predict 'fitness-to-fly' equally well in all patients. Patients at risk of hypercapnia with supplemental oxygen are not well studied. Th investigators will study children who have either neuromuscular weakness or central hypoventilation and who require nocturnal or intermittent daytime ventilator support.

The study also aims to assess feasibility of a randomised controlled trial (RCT) comparing the standard hypoxic standard test to a modified test designed to better suit children with type two respiratory failure.

DETAILED DESCRIPTION:
This study will assess feasibility of pulse oximetry (SpO2), end tidal carbon dioxide (ETCO2) and transcutaneous carbon dioxide partial pressure (TcCO2) measurement during a modified Hypoxic challenge test (HCT) in 12 children with neuromuscular weakness and 12 with central hypoventilation.

ELIGIBILITY:
Inclusion Criteria:

* ≤18 years
* Neuromuscular weakness or central hypoventilation
* Established nocturnal or intermittent daytime ventilatory support

Exclusion Criteria:

* Unable to sit in the plethysmograph
* Cardiac anomaly with right-to-left shunt

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
proof of concept outcome 1 | during hypoxic challenge test
  number of children/infants with SpO2 <90/85%
proof of concept outcome 2 | during hypoxic challenge test
  number of children with >15 mmHg rise in TcCO2/EtCO2

SECONDARY OUTCOMES:
Feasibility outcome 1: recruitment rate | one year
  recruitment rate
Feasibility outcome 2: protocol completion rate | one year
  protocol completion rate

CONTACTS AND LOCATIONS:
Overall Officials: Katharine C Pike, PhD, Principal Investigator — Great Ormond Street Hospital for Children NHS Foundation Trust
Locations (1):
- Great Ormond Street Hospital for Children NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided